CLINICAL TRIAL: NCT01235663
Title: Does Advisory Support to Prolong the Breast-feeding Period Reduce the Risk for Obesity and Metabolic Dysfunction in Infants of Obese Mothers ?
Brief Title: Minimizing the Risk for Obesity During Infancy by Extensive Advisory Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ole Pryds, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Breastfeeding-2650
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Reduce the Risk of Obesity During Infancy; Reduce the Risk of Insulin Resistance
Keywords: obesity, insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- advisory support (Experimental): advisory support for six months to prolong the breast-feeding period
  Interventions: Behavioral: advisory support

INTERVENTIONS:
Behavioral: advisory support — regular advisory support to the prolong breast-feeding period

SUMMARY:
0-hypothesis: advisory support does not

1. prolong the the breast-feeding period
2. minimize the risk of obesity and metabolic dysfunction in infants of obese mothers

ELIGIBILITY:
Inclusion Criteria:

Healthy, term infants Informed and written consent obtained from both parents -

Exclusion Criteria:

Sick infants Preterm infants No consent

-

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
fat tissue | 6 months
  weight skinfolds

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology, Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Carlsen EM, Kyhnaeb A, Renault KM, Cortes D, Michaelsen KF, Pryds O. Telephone-based support prolongs breastfeeding duration in obese women: a randomized trial. Am J Clin Nutr. 2013 Nov;98(5):1226-32. doi: 10.3945/ajcn.113.059600. Epub 2013 Sep 4. PMID 24004897